CLINICAL TRIAL: NCT06437327
Title: Comparison of Effectiveness Between Active Release Technique and Hold Relax Technique in Patients With Piriformis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/10
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Piriformis Syndrome
MeSH Terms: conditions — Piriformis Muscle Syndrome | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimiental Group 1 (Experimental): Hot pack for 10 minutes Interferential Current (IFC) for 10 minutes Active release technique is applied (patient is prone lying with knee flexed, Pressure is applied on taut band and patient is asked to move the leg in internal rotation to achieve maximal lengthening) Repetitions 5 to 7 times hold for 5 to 20 seconds
  Interventions: Procedure: Electrotherapy; Procedure: Active release technique
- Experimental Group 2 (Experimental): Hot pack for 10 minutes Interferential Current (IFC) for 10 minutes Hold relax technique This technique is applied while the patient is in supine lying with one leg crossed over the other Patient is instructed to contract the piriformis against the manual resistance for 5 to 10 secs Then 15 secs of passive stretch is given repetitions x 5 times
  Interventions: Procedure: Electrotherapy; Procedure: Hold relax technique

INTERVENTIONS:
Procedure: Electrotherapy — Hot pack for 10 minutes Interferential Current (IFC) for 10 minutes
Procedure: Active release technique — Active release technique is applied (patient is prone lying with knee flexed, Pressure is applied on taut band and patient is asked to move the leg in internal rotation to achieve maximal lengthening) Repetitions 5 to 7 times hold for 5 to 20 seconds
  Arms: Experimiental Group 1
Procedure: Hold relax technique — This technique is applied while the patient is in supine lying with one leg crossed over the other Patient is instructed to contract the piriformis against the manual resistance for 5 to 10 secs Then 15 secs of passive stretch is given repetitions x 5 times
  Arms: Experimental Group 2

SUMMARY:
This study is a randomized controlled trial and the purpose of this study is to compare the effects between active release technique and hold relax technique in patients with Piriformis syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effects between active release technique and hold relax technique in patients with piriformis syndrome pain, range of motion, and functional disability, in adults (age: 25-55 years)

1. Numeric pain rating scale
2. Goniometer
3. Oswestry Disability Questionairre Data will be collected before and after the intervention protocol for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post-intervention scores will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Gender: Both male and female
* Individuals aged 25-55 years
* Tenderness to palpation over sciatic foramen
* Positive FAIR Test.

Exclusion criteria :

* History of hip, pelvic, or Femoral fractures.
* Malignancies.
* Avascular necrosis of Femoral head.
* Inflammatory conditions (e.g. Rheumatoid Arthritis)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 2 weeks
  Numeric Pain Rating Scale (NPRS): ICC (0.93-0.96).It has a scale of 0-10 or 0-100 points and can be given verbally or in writing.
Physical Function using Oswestry disability Questionnaire | 2 weeks
  Physical Function will be measured using Oswestry disability Questionnaire
Hip internal rotation range of motion | 2 weeks
  Hip internal rotation using Goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan